CLINICAL TRIAL: NCT04647487
Title: EMBER-2: A Phase 1, Open-Label, Preoperative Window Study Evaluating the Biological Effects of LY3484356 in Post-menopausal Women With Stage I-III Estrogen Receptor-Positive, HER2-Negative Breast Cancer
Brief Title: A Study of LY3484356 in Women With Breast Cancer Before Having Surgery
Acronym: EMBER-2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 17575; J2J-MC-JZLB (Other: Eli Lilly and Company); 2020-002810-42 (EudraCT Number)
Record Dates: First submitted 2020-11-30; First posted 2020-12-01 (Actual); Results first posted 2025-11-12 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-10

CONDITIONS: Breast Cancer
Keywords: SERD
MeSH Terms: conditions — Breast Neoplasms | interventions — Imlunestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 200 milligrams (mg) LY3484356 (Experimental): Participants received 200 mg LY3484356 administered orally once daily for 15 days
  Interventions: Drug: LY3484356
- 400 mg LY3484356 (Experimental): Participants received 400 mg LY3484356 administered orally once daily for 15 days
  Interventions: Drug: LY3484356
- 800 mg LY3484356 (Experimental): Participants received 800 mg LY3484356 administered orally once daily for 15 days
  Interventions: Drug: LY3484356

INTERVENTIONS:
Drug: LY3484356 — Administered orally.
  Other Names: Imlunestrant

SUMMARY:
The purpose for this study is to see if the study drug, LY3484356, is safe and to determine what effects it has on breast cancer in participants with Estrogen Receptor Positive (ER+), HER2 Negative (HER2-) early stage (stage I-III) breast cancer, when given prior to surgery. Participation in this study could last up to 2.5 months.

ELIGIBILITY:
Inclusion Criteria:

* Have histologically confirmed invasive ER+, HER2- breast carcinoma
* Be willing and able to provide pre- and on-treatment tumor samples
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group scale
* Have adequate organ function
* Be able to swallow capsules
* Be a postmenopausal woman

Exclusion Criteria:

* Have bilateral invasive breast cancer
* Have metastatic breast cancer
* Plan to receive concurrent neoadjuvant therapy with any other non-protocol anti-cancer therapy
* Have had prior therapy (of any kind) for an invasive or non-invasive breast cancer
* Have had prior radiotherapy to the ipsilateral chest wall for any malignancy
* Have had prior anti-estrogen therapy with raloxifene, tamoxifen, aromatase inhibitor, or other selective estrogen receptor modulator (SERM), either for osteoporosis or prevention of breast cancer
* Have had prior hormone-replacement therapy within 4 weeks of the start of study treatment
* Have had major surgery within 28 days prior to randomization to allow for post-operative healing of the surgical wound and site(s)
* Have certain infections such as hepatitis or tuberculosis or HIV that are not well controlled
* Have another serious medical condition
* Have a history of any other cancer (except nonmelanoma skin cancer or carcinoma in-situ of the cervix), unless in complete remission with no therapy for a minimum of 3 years

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 87 (Actual)
Dates: Start 2021-04-21 (Actual); Primary Completion 2022-11-11 (Actual); Study Completion 2022-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (19):
- United States (8):
  - Winship Cancer Center Emory University, Atlanta, Georgia
  - Northwestern Memorial Hosptial, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Sarah Cannon Research Institute SCRI, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Vermont Medical Center, Burlington, Vermont
- Belgium (2):
  - Institut Jules Bordet, Brussel - Capital
  - Universitaire Ziekenhuizen Leuven - Campus Gasthuisberg, Leuven
- Hôpital René Huguenin, Saint-Cloud, Hauts-de-Seine, France
- Germany (3):
  - Universitätsklinikum Erlangen, Erlangen, Bavaria
  - Helios Kliniken Schwerin, Schwerin, Mecklenburg-Vorpommern
  - Klinikum der Universitaet Muenchen, München
- Spain (3):
  - Hospital Clinic I Provincial, Barcelona
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Madrid Norte Sanchinarro, Madrid
- United Kingdom (2):
  - The Royal Cornwall Hospital, Truro, Cornwall
  - Barts Cancer Institute, London, London City

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Study of LY3484356 in Women With Breast Cancer Before Having Surgery (EMBER-2) — https://trials.lillytrialguide.com/en-US/trial/3vEdhySNhh4bT91vRoma1P

RESULTS

PARTICIPANT FLOW:
Groups:
- 200 mg LY3484356: Participants received 200 mg LY3484356 administered orally once daily for 15 days
Period: Overall Study
Arm/Group | 200 mg LY3484356 | 400 mg LY3484356 | 800 mg LY3484356
Started | 28 | 30 | 29
Received At Least One Dose of Study Drug | 28 | 30 | 28
Completed (Participants who have completed all on-treatment visits were considered completers.) | 27 | 30 | 26
Not Completed | 1 | 0 | 3
Not completed — Protocol Deviation | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | 200 mg LY3484356 | 400 mg LY3484356 | 800 mg LY3484356 | Total
Number analyzed (Participants) | 28 | 30 | 28 | 86
Age, Continuous [Median (Full Range); unit: years] | 63.0 [50 to 74] | 63.5 [50 to 83] | 64.0 [50 to 83] | 63.5 [50 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 30 | 28 | 86
  Male | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 27 | 27 | 23 | 77
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 3 | 5 | 8
Region of Enrollment [Count of Participants; unit: Participants]
  Spain | 6 | 13 | 9 | 28
  Belgium | 6 | 6 | 7 | 19
  Germany | 5 | 7 | 6 | 18
  United States | 10 | 3 | 5 | 18
  France | 0 | 1 | 1 | 2
  United Kingdom | 1 | 0 | 0 | 1
Estrogen Receptor (ER) Expression [Mean (Standard Deviation); unit: H-score] — Tumor tissue collected by biopsy is used to determine ER expression. ER expression is measured by immunohistochemistry (IHC) and quantified by H-score. The H-score was calculated as the sum of multiplying the tumor cell ER staining intensity level 0 to 3 (0=none, 1=low, 2=moderate, 3=high) by the percentage (0 to 100) of cells at each intensity. Total ER H-score ranged from 0 to 300, where a higher score indicated stronger ER expression. Population: All enrolled participants with analyzable baseline and posttreatment data.
  H-score
    number analyzed (Participants) | 22 | 27 | 26 | 75
    (all) | 256.82 (42.33) | 289.81 (17.18) | 292.5 (13.36) | 281.07 (30.35)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Estrogen Receptor (ER) Expression
Description: Tumor tissue collected by biopsy is used to determine ER expression. ER expression is measured by immunohistochemistry (IHC) and quantified by H-score. The H-score was calculated as the sum of multiplying the tumor cell ER staining intensity level 0 to 3 (0=none, 1=low, 2=moderate, 3=high) by the percentage (0 to 100) of cells at each intensity. Total ER H-score ranged from 0 to 300, where a higher score indicated stronger ER expression. Percent change in ER expression was defined as 100*(ER expression on-treatment - ER expression pre-treatment)/(ER expression pre-treatment). Geometric mean percent change and 90 percent (%) confidence interval for percent change were obtained from a t-test of the log ratio i.e. log(ER expression on-treatment/ER expression pre-treatment).
Time Frame: Baseline, Day 15
Population: All enrolled participants with analyzable baseline and posttreatment data.
Measure: Geometric Mean (90% Confidence Interval); unit: percent change
Arm/Group | 200 mg LY3484356 | 400 mg LY3484356 | 800 mg LY3484356
Number analyzed (Participants) | 22 | 27 | 26
percent change | -88.89 [-95.62 to -71.85] | -81.50 [-91.34 to -60.47] | -70.13 [-78.38 to -58.75]

2. Secondary Outcome: Percent Change From Baseline in Ki-67
Description: Tumor tissue collected by biopsy is used to determine Ki-67 expression. It is measured by IHC and the Ki-67 index is defined as the percent of cells staining positive by validated central assay. Percent change in Ki-67 index was defined as 100*(Ki-67 index on-treatment - Ki-67 index pre-treatment)/(Ki-67 index pre-treatment). Geometric mean percent change and 90 percent (%) confidence interval for percent change were obtained from a t-test of the log ratio i.e. log(Ki-67 index on-treatment/Ki-67 index pre-treatment).
Time Frame: Baseline, Day 15
Population: All enrolled participants with analyzable baseline and posttreatment data.
Measure: Geometric Mean (90% Confidence Interval); unit: percent change
Arm/Group | 200 mg LY3484356 | 400 mg LY3484356 | 800 mg LY3484356
Number analyzed (Participants) | 21 | 22 | 20
percent change | -68.56 [-78.71 to -53.59] | -70.61 [-80.04 to -56.73] | -72.28 [-81.22 to -59.09]

3. Secondary Outcome: Percent Change From Baseline in Progesterone Receptor (PR) Expression
Description: Tumor tissue collected by biopsy is used to determine PR expression. PR expression is measured by IHC and quantified by H-score. The H-score was calculated as the sum of multiplying the tumor cell ER staining intensity level 0 to 3 (0=none, 1=low, 2=moderate, 3=high) by the percentage (0 to 100) of cells at each intensity. Total PR H-score ranged from 0 to 300, where a higher score indicated stronger PR expression. Percent change in PR expression was defined as 100*(PR expression on-treatment - PR expression pre-treatment)/(PR expression pre-treatment). Geometric mean percent change and 90 percent (%) confidence interval for percent change were obtained from a t-test of the log ratio i.e. log(PR expression on-treatment/PR expression pre-treatment).
Time Frame: Baseline, Day 15
Population: All enrolled participants with analyzable baseline and posttreatment data.
Measure: Geometric Mean (90% Confidence Interval); unit: percent change
Arm/Group | 200 mg LY3484356 | 400 mg LY3484356 | 800 mg LY3484356
Number analyzed (Participants) | 20 | 26 | 26
percent change | -85.44 [-96.61 to -37.36] | -75.56 [-90.33 to -38.20] | -82.01 [-91.98 to -59.66]

4. Secondary Outcome: Pharmacokinetics (PK): Plasma Concentration of LY3484356
Description: Plasma Concentration of LY3484356 evaluated using sparse sampling methodology
Time Frame: Day 1: 3.5 hours (h) postdose; Day 8: Predose; Day 8: 3.5 h postdose
Population: All enrolled participants who received at least one full dose of study drug and have at least one postbaseline evaluable PK sample.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliter (ng/mL)
Arm/Group | 200 mg LY3484356 | 400 mg LY3484356 | 800 mg LY3484356
Number analyzed (Participants) | 27 | 27 | 25
nanograms/milliliter (ng/mL)
  Day 1 (3.5 h Postdose) | 25.3 (74) | 86.9 (82) | 106 (107)
  Day 8 (Predose) | 33.0 (70) | 74.3 (77) | 99.6 (87)
  Day 8 (3.5 h Postdose) | 55.2 (58) | 120 (63) | 225 (77)

ADVERSE EVENTS:
Time Frame: Baseline until end of follow-up (up to 63 days)
Description: All enrolled participants who received at least one dose of study drug.
Arm/Group | 200 mg LY3484356 | 400 mg LY3484356 | 800 mg LY3484356
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/30 | 0/28
Serious Adverse Events (participants affected / at risk) | 1/28 | 2/30 | 1/28
Other Adverse Events (participants affected / at risk) | 15/28 | 12/30 | 15/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 200 mg LY3484356 (N=28) | 400 mg LY3484356 (N=30) | 800 mg LY3484356 (N=28)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Mastitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 200 mg LY3484356 (N=28) | 400 mg LY3484356 (N=30) | 800 mg LY3484356 (N=28)
Leukopenia (Blood and lymphatic system disorders) | 3 (4) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (4) | 3 (3) | 9 (9)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1) | 4 (4)
Asthenia (General disorders) | 0 (0) | 4 (4) | 1 (1)
Fatigue (General disorders) | 2 (2) | 2 (2) | 3 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (3)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 2 (2) | 2 (4)
Breast pain (Reproductive system and breast disorders) | 2 (4) | 2 (2) | 2 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 4 (4) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2022-01-18): https://cdn.clinicaltrials.gov/large-docs/87/NCT04647487/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-09): https://cdn.clinicaltrials.gov/large-docs/87/NCT04647487/SAP_001.pdf